CLINICAL TRIAL: NCT07036692
Title: The FaibaGo Study - Long-Term Weight Reduction Via Low-Threshold Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: DCB Research AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FaibaGo
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Nutritional and Metabolic Diseases; Overweight
Keywords: Overweight; Chewing gum; Galactooligosaccharides; GOS (Galactooligosaccharides); Oral microbiome; Intestinal microbiome
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Chewing gum containing maltitol powder
  Interventions: Dietary Supplement: Placebo
- Interventional (Experimental): Chewing gums containing galactooligosaccharides (GOS)
  Interventions: Dietary Supplement: FibreGum
- No-treatment control (No Intervention): No chewing-gums

INTERVENTIONS:
Dietary Supplement: Placebo — To chew every day during a period of 4 months 3 chewing gums (morning, noon and evening) for at least 20 minutes each.
  Arms: Placebo
Dietary Supplement: FibreGum — To chew every day during a period of 4 months 3 chewing gums (morning, noon and evening) for at least 20 minutes each.
  Arms: Interventional

SUMMARY:
The main aim of this study is to assess the effect of a chewing gum containing galactooligosaccharides (GOS) on the body mass index (BMI), the metabolism and the oral and intestinal microbiomes in a population of overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent (IC) according to ICH/GCP regulations prior to any study-specific procedures
* Adults aged ≥ 25 years
* Overweight as determined by a Body Mass Index > 25 kg/m2
* Metabolic risk factor: at least one of the following criteria:

  i. HbA1c ≥ 5.7% ii. Elevated liver enzymes (ALAT, ASAT, Gamma-Glutamyltransferase (gGT) at least one above normal range of the assay used in the respective laboratory) iii. LDL-cholesterol > 3.0 mmol/l iv. Triglycerides > 1.7 mmol/l
* Ability and willingness to follow the study protocol (e.g., cognitive capacity for compliance, gum chewing, faecal sample collection)
* Access to a scale to self-report weight
* Access and willing to use an electronic device (e.g., mobile phone, computer or tablet)
* Laboratory assessments of blood parameters were performed within a reasonable timeframe prior to the eligibility assessment, as determined by the PI.

Exclusion Criteria:

* Systemic antibiotic use within the last 2 months
* History of bariatric surgery
* Initiation or dose adjustment of pharmaceutical treatment for dyslipidemia or hyperglycemia within the last 3 months or during the study (e.g., metformin, statins, SGLT2 inhibitors)
* Use of prebiotic or probiotic supplementation (duration >1 month) within the last 6 weeks (at PI's discretion, based on medication summary of TP)
* Medical weight management treatments within the last year (e.g., Glucagon-Like Peptide-1 (GLP-1) agonists)
* Recent (<1 month) dose adjustment, initiation or termination of proton pump inhibitors use (e.g., pantoprazole, omeprazole)
* Professionally supervised intensive (>6 months of ongoing supervision) weight management treatments (e.g., structured nutrition counselling) within the last year (at the PI's discretion)
* Diagnosis of Type 1 or Type 2 diabetes requiring bolus insulin therapy or frequent dose adjustments in base line insulin
* Regular alcohol consumption exceeding two (women) or three (men) standard units (10 g of pure alcohol) per day
* Consumption of more than one nicotine product (e.g., (e-)cigarette, gum) per month
* Regular drug abuse (once per week over the past 4 months)
* Any stage of known pregnancy or lactation period (self-reported)
* Active cancer or recent cancer treatment (within the last 4 months)
* Chronic, active inflammatory diseases (e.g., inflammatory bowel disease, rheumatoid arthritis)
* Severe gastrointestinal disorders (e.g., celiac disease, short bowel syndrome, gastroparesis)
* Known eating disorder (medically diagnosed)
* Participation in another investigation with an investigational drug within the 30 days preceding randomisation
* Dependency from the Sponsor-Investigator
* Last visit with TP > 22 days prior to eligibility assessment

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Body Mass Index (BMI) during intervention | 4 months
  Difference in the BMI measured at intervention start and intervention completion

SECONDARY OUTCOMES:
Systolic blood pressures change during intervention | 4 months
  Difference in systolic blood pressure (mm Hg) between intervention completion and intervention start.
Diastolic blood pressures changes during intervention | 4 months
  Difference in diastolic blood pressure (mm Hg) between intervention completion and intervention start.
Self-reported weight changes during intervention | 4 months
  Difference in self-reported weight (kg) between intervention completion and intervention start.
Self-reported weight changes during follow-up | 2 months from intervention completion (month 4) to end of follow-up period (month 6)
  Difference in self-reported weight (kg) between end of follow-up period and intervention completion.
Waist circumference changes during intervention | 4 months
  Difference in waist circumference (cm) between between intervention completion and intervention start.
Waist circumference changes during follow-up | 2 months from intervention completion (month 4) to end of follow-up period (month 6)
  Difference in waist circumference (cm) between end of follow-up period and intervention completion.
Fasting blood glucose change during intervention | 4 months
  Difference in fasting blood glucose (mg/dL or mmol/L) between intervention completion and intervention start.
Fasting insulin change during intervention | 4 months
  Difference in fasting insulin (mIU/mL) between intervention completion and intervention start.
HOmeostatic Model Assessment of Insulin Resistance (HOMA-IR) index change during intervention | 4 months
  Difference in Homeostatic Model Assessment of Insulin Resistance Index (min:0 - max:10) between intervention completion and intervention start. Lower scores mean better outcome.
Hemoglobin A1c (HbA1c) change during intervention | 4 months
  Difference in HbA1c (mmol/mol) between intervention completion and intervention start.
Cholesterol change during intervention | 4 months
  Difference in Cholesterol (mg/dL) between intervention completion and intervention start.
Triglyceride change during intervention | 4 months
  Difference in Triglyceride (mg/dL) between intervention completion and intervention start.
High-density lipoproteins (HDL) change during intervention | 4 months
  Difference in HDL (mg/dL) between intervention completion and intervention start.
Low-density lipoproteins (LDL) change during intervention | 4 months
  Difference in LDL (mg/dL) between intervention completion and intervention start.
Neutrophils change during intervention | 4 months
  Difference in Neutrophils count (%) between intervention completion and intervention start.
Lymphocytes change during intervention | 4 months
  Difference in Lymphocytes count (%) between intervention completion and intervention start.
Monocyte change during intervention | 4 months
  Difference in Monocytes count (%) between intervention completion and intervention start.
Eosinophils change during intervention | 4 months
  Difference in Eosinophils count (%) between intervention completion and intervention start.
Basophils change during intervention | 4 months
  Difference in Basophils count (%) between intervention completion and intervention start.
Alanine Aminotransferase (ALAT) change during intervention | 4 months
  Difference in ALAT (U/L) between intervention completion and intervention start.
Aspartate Aminotransferase (ASAT) change during intervention | 4 months
  Difference in ASAT (U/L) between intervention completion and intervention start.
Calcifediol (25OH-Vitamin D3) change during intervention | 4 months
  Difference in Calcifediol (nmol/L) between intervention completion and intervention start.
Thyroid-Stimulating Hormone (TSH) change during intervention | 4 months
  Difference in TSH (mU/L) between intervention completion and intervention start.
Ferritin change during intervention | 4 months
  Difference in Ferritin (μg/L) between intervention completion and intervention start.
Proteinuria change during intervention | 4 months
  Difference in Proteinuria (g/24h) between intervention completion and intervention start.
Oral microbiome change during intervention | 4 months
  Change in oral microbiota as assessed by metagenomic sequencing from oral washes between intervention completion and intervention start.
Gut microbiome change during intervention | 4 months
  Change in intestinal microbiota-composition as assessed by metagenomic sequencing from stool samples between intervention completion and intervention start.
Breath metabolome change during intervention | 4 months
  Change in volatile compounds present in the breath detected by secondary electrospray ionization (SESI) source in combination with a high-resolution mass spectrometry (HR-MS) between intervention completion and intervention start.
Body composition change (body fat) during intervention | 4 months
  Change in body fat between intervention completion and intervention start.
Body composition change (lean mass) during intervention | 4 months
  Change in lean mass between intervention completion and intervention start.
Change in in-vitro response of faecal microbiota (alpha diversity) to a panel of prebiotic compounds during intervention | 4 months
  Change in community diversity (alpha diversity) assessed by metagenomic sequencing between intervention completion and intervention start.
Change in in-vitro response of faecal microbiota (beta diversity) to a panel of prebiotic compounds during intervention | 4 months
  Change in composition (beta diversity, differential abundance) assessed by metagenomic sequencing between intervention completion and intervention start.

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Balmer, Prof. med., Principal Investigator — Department of Biomedical Research, University of Bern
Locations (1):
- Department of Biomedical Research, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No